CLINICAL TRIAL: NCT04017507
Title: The Effects of Oscillating-Rotating Electric Toothbrushes on Plaque and Gingival Health: A Meta-Analysis
Brief Title: The Effects of Oscillating-Rotating Electric Toothbrushes on Plaque and Gingival Health
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019BrushMetaAnalysis
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Gingivitis; Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oscillating-rotating electric toothbrush: Twice daily brushing
  Interventions: Device: Oscillating-rotating electric toothbrush
- Side-to-side electric toothbrush: Twice daily brushing
  Interventions: Device: Side-to-side electric toothbrush
- Manual toothbrush: Twice daily brushing
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Oscillating-rotating electric toothbrush — Oscillating-rotating electric toothbrush used twice daily
  Groups: Oscillating-rotating electric toothbrush
Device: Side-to-side electric toothbrush — Side-to-side electric toothbrush used twice daily
  Groups: Side-to-side electric toothbrush
Device: Manual toothbrush — Manual toothbrush used twice daily
  Groups: Manual toothbrush

SUMMARY:
The aim of this analysis was to compare the effects of oscillating-rotating (O-R), side-to-side (sonic), and manual toothbrushes on plaque and gingival health after multiple uses.

ELIGIBILITY:
Subjects were excluded from this study for the following reasons;

* pregnancy,
* rampant caries,
* severe periodontitis,
* at discretionary of the Principal Investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This meta-analysis includes healthy adult male and females.
Sampling Method: Probability Sample
Enrollment: 2145 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Bleeding Sites | Up to 12 weeks
  Change from baseline as measured on number of bleeding sites ( via gingival bleeding index, Loe Silness index, Papillary bleeding index or Mazza gingival index).
Dental Plaque Scores | Up to 12 weeks
  Change from baseline as measured by mean plaque score reduction from baseline (via Turesky's Modification of Quigley-Hein index, or Rustogi Modified Navy Plaque Index).

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple P&G Investigation Clinical Sites, Cincinnati, Ohio, United States